CLINICAL TRIAL: NCT03717142
Title: Feasibility of the LUM Imaging System for in Vivo and Ex Vivo Detection of Cancer in Subjects with Low Grade Gliomas, Glioblastomas, and Cancer Metastases to the Brain
Brief Title: Feasibility of the LUM Imaging System for Detection of Cancer to the Brain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Initial data indicated a change in study design required prior to collecting additional data.
Sponsor: Lumicell, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: CL0004
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-03

CONDITIONS: Low Grade Glioma of Brain; Glioblastoma; Metastasis to Brain
Keywords: Fluorescence; Brain; Cancer detection
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Dose Escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Auto-fluorescence (No Intervention): No LUM015 injection will be given to three (3) patients, in each indication, to measure baseline tissue fluorescence. Imaging with the LUM imaging device will be performed in vivo and ex vivo on surgical tissue.
- 1st Tier Dose Level (Experimental): 3 patients, in each indication, will be administered a single dose of LUM015 at 1.0 mg/kg.Imaging with the LUM imaging device will be performed in vivo and ex vivo on surgical tissue.
  Interventions: Combination Product: LUM Imaging System
- 2nd Tier Dose Level (Experimental): 3 patients, in each indication, will be administered a single dose of LUM015 at 2.0 mg/kg. Imaging with the LUM imaging device will be performed in vivo and ex vivo on surgical tissue.
  Interventions: Combination Product: LUM Imaging System
- 3rd Tier Dose Level (Experimental): After an interim analysis, the dosing for the 3 patients, in each indication, will be administered a single dose of LUM015 of no greater than 3.0 mg/kg. Imaging with the LUM imaging device will be performed in vivo and ex vivo on surgical tissue.
  Interventions: Combination Product: LUM Imaging System

INTERVENTIONS:
Combination Product: LUM Imaging System — Patients will be injected with one of 3 study doses of LUM015, or have no LUM015 intervention, and tissue will be imaged in vivo and ex vivo with the LUM imaging device.
  Arms: 1st Tier Dose Level; 2nd Tier Dose Level; 3rd Tier Dose Level

SUMMARY:
The overall objective of this study is to assess the safety and efficacy of the LUM Imaging System in imaging primary and metastatic cancer in the brain. This includes selecting a dose to determine the initial efficacy of LUM015 for the molecular imaging of low-grade gliomas, glioblastomas and cancer masses that have metastasized to the brain.

DETAILED DESCRIPTION:
The primary objective of this feasibility study is to identify an effective dose of LUM015 for imaging low grade gliomas, glioblastomas and cancer metastases to the brain. The optimal dose will be used for future studies. Both normal brain tissue and tumor tissue will be imaged and analyzed using the LUM Imaging device. The LUM Imaging System is a combination product consisting of the LUM Imaging Device and the imaging agent LUM015.

Subjects with a possible diagnosis of low grade glioma, glioblastoma and metastases to the brain, and scheduled for surgical resection, will be screened, recruited. On day of scheduled surgery, the subject will be administered with LUM015 4 ± 2 hours prior to using LUM Imaging System during surgery. LUM015 will be administered via peripheral intravenous (IV) injection as a single dose between 1.0 - 3.0 mg/kg.

Before the tumor mass is resected, the LUM Imaging Device will be used to scan images of distinct areas of grossly normal appearing brain tissue and, separately, images of distinct areas of grossly appearing tumor. Following tumor mass resection, the tumor bed is scanned to record in vivo images. The resected tissue will also be imaged ex vivo.

All subjects will continue to be monitored until hospital discharge and followed through their first standard of care post-surgical visit. Subjects with adverse events that are determined to be possibly related to the investigational product will continue to be followed until resolution or stabilization of the adverse event.

ELIGIBILITY:
Inclusion Criteria:

* Has radiologic imaging with a presumed diagnosis of low grade gliomas, glioblastoma/ grade III glioma or cancer metastases to the brain and must be scheduled for surgical resection
* Male or female subjects 18 years of age or older
* Subjects must have normal liver, kidney, and bone marrow function as defined below:

  * Leukocytes > 3,000/mcL
  * Platelets > 100,000/mcL
  * total bilirubin within normal institutional limits
  * AST (SGOT)/ALT (SGPT) < 2.5 X institutional upper limit of normal
  * Creatinine ≤ 1.5 mg/dL or creatinine clearance > 60 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal.
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) starting the day entering the study, and for 60 days after injection of the imaging agent
* Subjects with ECOG performance status of 0 or 1

Exclusion Criteria:

* Subjects previously treated with systemic therapies to treat the cancer to be removed during this clinical investigation, such as neo-adjuvant chemotherapy or hormonal therapy.
* Subjects with a known current condition of substance addiction.
* Subjects who have taken an investigational drug within 30 days of enrollment or those who have not recovered from adverse events due to pharmaceutical or diagnostic agents.
* Subjects with uncontrolled hypertension defined as persistent systolic blood pressure > 180 mm Hg, or diastolic blood pressure > 110 mm Hg; those subjects with known HTN should be stable within these ranges while under pharmaceutical therapy.
* History of allergic reaction attributed to drugs containing polyethylene glycol (PEG).
* History of allergic reaction to any oral or intravenous contrast agents.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, COPD or asthma requiring hospitalization within the past 12 months, or psychiatric illness/social situations that would limit compliance with study requirements.
* Subjects who are pregnant or nursing.
* Subjects who are sexually active and not willing/able to use medically acceptable forms of contraception upon entering the study.
* HIV-positive individuals on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with LUM015.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
Correlation of fluorescence levels in normal and tumor tissue by dose of LUM015 | Day 1
  Correlate the fluorescence levels in normal and tumor tissue from specimen imaging to the dose of LUM015 injected, or if not injected. Determine initial efficacy of LUM015 in labeling primary and metastatic cancer in the Brain by molecular imaging compared with imaging results in pathology.

SECONDARY OUTCOMES:
Number of reported safety events | up to 14 days post surgery
  Reported adverse events will be assessed and aggregated according to event type, relation to device or drug, and severity

CONTACTS AND LOCATIONS:
Overall Officials: E. Antonio Chiocca, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided